CLINICAL TRIAL: NCT04651530
Title: Endoscopic Cyclophotocoagulation in Normal Tension Glaucoma
Acronym: ECPNTG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Prof. Mika Harju, Head of Glaucoma department, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 876543
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Normal Tension Glaucoma; Cataract
Keywords: endoscopic cyclophotocoagulation; ECP; Surgery
MeSH Terms: conditions — Low Tension Glaucoma; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phaco (Active Comparator): Cataract surgery only
  Interventions: Procedure: Phaco
- Phaco+ECP (Experimental): Cataract surgery combined with endoscopic cyclophotocoagulation
  Interventions: Procedure: Phaco+ECP

INTERVENTIONS:
Procedure: Phaco — phacoemulsification of cataract only
  Arms: Phaco
Procedure: Phaco+ECP — Endoscopic cyclophotocoagulation is done in the same procedure as phacoemulsification of cataract
  Arms: Phaco+ECP

SUMMARY:
The purpose of this study is to assess whether endoscopic cyclophotocoagulation added to cataract surgery lowers intraocular pressure more than cataract surgery alone in patients with normal tension glaucoma.

DETAILED DESCRIPTION:
Subjects with normal tension glaucoma that is stable with current medication needing cataract surgery are recruited in the study. All patients meeting the inclusion criteria and giving informed consent will be randomized to whether having endoscopic cyclophotocoagulation performed in the same session with cataract surgery, or cataract surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Normal Tension Glaucoma with typical nerve fiber layer defects in red-free photographs and/or optical coherence tomography (OCT) and possible equivalent visual field defects, IOP never more than 21 mmHg, and open anterior chamber angle
* Glaucoma stable with current medication assessed by a glaucoma specialist
* Clinically significant cataract

Exclusion Criteria:

* Secondary Glaucoma e.g. due to previous injury or uveitis
* Exfoliation syndrome
* Pigment dispersion syndrome
* Previous transscleral or endoscopic cyclophotocoagulation
* Previous other glaucoma surgery
* Cataract due to eye injury or congenital cataract
* Zonular weakness due to Marfan syndrome or other
* Previous retinal detachment
* Previous intraocular surgery like vitrectomy and other retinal surgery
* Wet age-related macular degeneration
* Diabetic retonopathy
* Previous corneal transplant or previous refractive surgery
* Fuchs' dystrophy and other abnormalities compromising corneal clarity like scars
* The patient does not want to participate in the study
* The glaucoma progresses on current IOP
* The patient does not speak Finnish, Swedish or English
* Dementia
* Only eye with vision worse than 20/200 or loss of central visual field

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Succes rate | One year postoperatively
  Success: Decrease in Intraocular Pressure (IOP) of 20 % or more or former level with fewer medications

SECONDARY OUTCOMES:
Additional surgery | Five years postoperatively
  Comparison of the need for additional glaucoma surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mika Harju, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland